CLINICAL TRIAL: NCT04992637
Title: ClockWork: Harnessing the Circadian Timing System for Postpartum Weight Management & Health
Brief Title: ClockWork Postpartum Weight Management Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: The Obesity Society (Other); WW International Inc (Industry)
Responsible Party: Principal Investigator, Rachel Kolko, Research Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19120236
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Obesity; Postpartum Weight Retention; Weight Gain, Maternal
MeSH Terms: conditions — Obesity; Gestational Weight Gain | interventions — Cwo protein, Drosophila

STUDY DESIGN:
Intervention Model Description: Women will be randomized to receive either the ClockWork intervention or Usual Care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ClockWork (Experimental): Participants who are randomized to treatment will receive the ClockWork intervention
  Interventions: Behavioral: ClockWork
- Usual Care (Active Comparator): Participants will receive usual care during the postpartum period.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: ClockWork — ClockWork is a behavioral weight loss intervention comprised of coaching sessions as well as digital monitoring and feedback tools. It addresses 4 key behaviors related to the CTS, weight, and health and their Amount, Regularity & Timing-the ART of ClockWork. Women will receive 12 tailored coaching sessions to review their digital monitoring of each key behavior, learn intervention content, and set goals, which are delivered in-person, by phone, or web to fit women's needs postpartum. Coaches will use women's baseline responses to tailor sessions around the key behaviors. The investigators will protocolize real-time monitoring to increase engagement and adherence, and to facilitate just-in-time adaptive reminders, recommendations, and coaching sessions.
  Arms: ClockWork
Other: Usual Care — Usual Care consists of the standard care that postpartum women receive without any additional intervention components.
  Arms: Usual Care

SUMMARY:
The ClockWork Postpartum Weight Management Pilot Study is an intervention study that will assess the feasibility, acceptability, and initial efficacy of the ClockWork intervention among women with prepregnancy overweight/obesity during the first 4 months postpartum.

DETAILED DESCRIPTION:
Overview of Procedures. The investigators developed a prototype mobile app to monitor ClockWork target behaviors, and now aim to gain stakeholder input to refine the interface and improve usability via feedback from postpartum women who began pregnancy with obesity. In this pilot trial, women will complete baseline assessments in the first month postpartum and be randomized to either usual care or ClockWork for 4 months, then complete assessments.

Participants & Recruitment. Given that the investigators want to initiate treatment quickly after delivery, women will be recruited at the end of pregnancy through Magee-Womens Hospital. Women will be randomized to receive either the ClockWork intervention or Usual Care. ClockWork is a behavioral weight loss intervention comprised of coaching sessions as well as digital monitoring and feedback tools. It addresses 4 key behaviors related to the circadian timing system (CTS), weight, and health and their Amount, Regularity & Timing-the ART of ClockWork. Women will receive 12 tailored coaching sessions to review digital monitoring of each key behavior, learn intervention content, and set goals, which are delivered in-person, by phone, or web to fit women's needs postpartum. Coaches (Dr. Kolko Conlon or study interventionist) will use women's baseline responses to tailor sessions around the key behaviors. The investigators will protocolize real-time monitoring to increase engagement and adherence, and to facilitate just-in-time adaptive reminders, recommendations, and coaching sessions. Usual Care does not involve any additional intervention.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Prenatal BMI greater than or equal to 25
* At least 28 weeks gestation
* English speaking
* Singleton pregnancy

Exclusion Criteria:

* Preexisting diabetes
* Use of medications known to affect weight (example, second generation antipsychotics)
* Enrolled in current weight management programming
* Recent weight loss surgery (within the past 3 years)
* Women who endorse acute psychiatric symptoms (e.g., suicidality) that warrant immediate treatment will be excluded and referred for care.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of sessions attended among women randomized to receive the ClockWork Intervention | First 4 months postpartum
  Number of sessions attended will be calculated for each participant
The percentage of days with completed monitoring among women randomized to receive the ClockWork Intervention | First 4 months postpartum
  Women will be asked to monitor daily
Participant liking of ClockWork (sessions, content, digital monitoring interface) | First 4 months postpartum
  Participant liking will be assessed using a Program Evaluation measure designed for this study. The measure uses a 10-point Likert Scale ranging from "not at all" (1) to "a lot" (10). Higher scores on this measure indicate greater satisfaction with ClockWork program components.
Perceived utility ratings of ClockWork (sessions, content, digital monitoring interface) | First 4 months postpartum
  Perceived utility will be assessed using a Program Evaluation measure designed for this study. The measure uses a 10-point Likert Scale ranging from "not helpful at all" (1) to "extremely helpful" (10). Higher scores on this measure indicate greater satisfaction with ClockWork program components.
Changes in the "ART" (amount, regularity, and timing of targeted intervention behaviors) from baseline to 4 months postpartum | First 4 months postpartum
  A composite score will be calculated to assess changes in the "ART" of behaviors. Participants will record the "ART" of targeted intervention behaviors using self-monitoring forms designed for the study.
Weight change from delivery to 4 months postpartum | First 4 months postpartum
  Weight in lbs.
Weight change from prepregnancy to 4 months postpartum | Pre-pregnancy through 4 months postpartum
  Weight in lbs.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Kolko, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No